CLINICAL TRIAL: NCT03619135
Title: Effectiveness of External Vibration for Pain Relief During Peripheral Intravenous Cannulation in Adult Patients
Brief Title: Effectiveness of External Vibration for Pain Relief During Intravenous Access in Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyle Stein (Other)
Responsible Party: Sponsor-Investigator, Kyle Stein, Principal Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201601806
Record Dates: First submitted 2018-08-02; First posted 2018-08-07 (Actual); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Pain Management; Anxiety
Keywords: Pain; Anxiety; intravenous access
MeSH Terms: conditions — Agnosia; Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Use of Buzzy Device (Experimental): The Buzzy device was used for IV access for this arm.
  Interventions: Device: Buzzy
- Control (Placebo Comparator): No Buzzy device was used - standard IV access for this arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Buzzy — The Buzzy is a reusable device that applies vibration to the skin surface to override the body's gate control pain pathway. It has been used effectively to reduce the discomfort of intravenous cannulation (IV placement) in pediatric patients. Also, it has been utilized to reduce the discomfort of injections in pediatric and adult patients. We are preforming this study to evaluate the effectiveness of the Buzzy in reducing the discomfort associated with intravenous cannluation (IV placement) in adults.
  Arms: Use of Buzzy Device
Other: Placebo — No use of the Buzzy (standard IV access techniques)
  Arms: Control

SUMMARY:
A large number of dentoalveolar (tooth extraction) procedures performed by Oral and Maxillofacial Surgeons utilize intravenous sedation. Procedures commonly performed may include surgical removal of teeth, bone grafting, surgical placement of dental implants, and removal of cysts or tumors from the jaws, among others. Obtaining peripheral intravevenous (IV) cannulation often proves to be a very stressful and anxious event for the patient. The anxiety and stress from the venipuncture alone affects not only the psychological stability of the patient, but also the patient's physiology. The Buzzy vibration external stimulation device has shown to be an effective tool in pediatric venipunture procedures. The aim of this study is to investigate the effects of the Buzzy stimulation device in pain and anxiety reduction during peripheral intravenous cannulation in an adult population.

Enrollees in this study will be patients who will undergo dental surgery with intravenous sedation. The patients who are enrolled will receive an IV either with or without the Buzzy. The Buzzy is a small vibration device which will be placed next to the IV placement site.

DETAILED DESCRIPTION:
The participants will be randomized into two groups, those who use the Buzzy system (experimental), and routine IV start (control). Prior to knowing their group, all patients will answer the "Before Intravenous Catheterization" portion of the form in order to eliminate bias. After this portion is complete, their group (experimental vs control) will be determined from opening a blinded envelope.

A tourniquet will be placed, followed by the Buzzy stimulation device (if in the experimental group). An alcohol swab will be used and then a 22 gauge IV catheter will be inserted, connected to fluids, and secured with tape. The antecubital fossa or the dorsal hand/wrist will be the only sites used in the study. All participants will fill out the post-insertion questions on the form and those patients that used the Buzzy system will then fill out the several specific questions related to the experimental group. This will conclude the patient's involvement in the study. The patient will then continue with treatment as planned. We will plan to exclude cases where the IV is not obtained on the first attempt, if a smaller or larger gauge IV catheter is required, or if an insertion site not listed above is required. The case will be excluded if adjunctive steps are taken to obtain IV access (i.e. Oral sedation, nitrous oxide, heat packs).

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and 40.
* Eligible for third molar removal with sedation.

Exclusion Criteria:

* Not eligible for surgery.
* Not eligible for sedation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2017-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle M Stein, DDS, FACS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa College of Dentistry, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canbulat N, Ayhan F, Inal S. Effectiveness of external cold and vibration for procedural pain relief during peripheral intravenous cannulation in pediatric patients. Pain Manag Nurs. 2015 Feb;16(1):33-9. doi: 10.1016/j.pmn.2014.03.003. Epub 2014 Jun 7. PMID 24912740
- [Background] Inal S, Kelleci M. Relief of pain during blood specimen collection in pediatric patients. MCN Am J Matern Child Nurs. 2012 Sep;37(5):339-45. doi: 10.1097/NMC.0b013e31825a8aa5. PMID 22895207
- [Background] Baxter AL, Cohen LL, McElvery HL, Lawson ML, von Baeyer CL. An integration of vibration and cold relieves venipuncture pain in a pediatric emergency department. Pediatr Emerg Care. 2011 Dec;27(12):1151-6. doi: 10.1097/PEC.0b013e318237ace4. PMID 22134226

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Use of Buzzy Device | Control
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Use of Buzzy Device | Control | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 26 | 55
  Male | 21 | 24 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain
Description: Pain is measured on a 10 point visual analog scale with 0 being no pain and 10 being the worst pain imaginable. A higher score is a worse outcome.
Time Frame: Baseline and after IV access
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Use of Buzzy Device | Control
Number analyzed (Participants) | 50 | 50
score on a scale | 1.55 (1.119) | 1.76 (1.401)

2. Primary Outcome: Change in Anxiety
Description: Anxiety is measured on a 10 point visual analog scale with 0 being no anxiety and 10 being the worst anxiety imaginable. A higher score is a worse outcome.
Time Frame: Baseline and after IV access
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Use of Buzzy Device | Control
Number analyzed (Participants) | 50 | 50
score on a scale | 1.70 (1.743) | 1.84 (1.796)

ADVERSE EVENTS:
Time Frame: The entirety of the study for each patient. This was approximately 5 minutes for the IV access (portion involving the research) and approximately 60 minutes for the total surgical procedure.
Description: No adverse events were encountered.
Arm/Group | Use of Buzzy Device | Control
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT03619135/Prot_SAP_000.pdf